CLINICAL TRIAL: NCT02955147
Title: Open Label Study to Test the Safety and Efficacy of Ustekinumab in Patients With Giant Cell Arteritis
Brief Title: Ustekinumab for the Treatment of Giant Cell Arteritis
Acronym: UGCA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inefficacy
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sebastian H Unizony, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000932
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Giant Cell Arteritis; Temporal Arteritis; Horton's Disease
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Ustekinumab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ustekinumab plus prednisone (Experimental): 1. Ustekinumab: 90 mg of ustekinumab will be administered subcutaneously at baseline, week 4, week 12, week 20, week 28, week 36 and week 44.
  2. Prednisone: All patients will receive a prednisone course tapered according to predefined schedules starting at either 60 mg, 40 mg or 20 mg. The initial dose of prednisone will be chosen by the investigators according to disease severity and comorbid medical conditions. The duration of the prednisone taper will be 6 months in all cases.
  Interventions: Drug: Ustekinumab; Drug: Prednisone

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab is a humanized monoclonal antibody that targets the p40 subunit of IL-12 and IL-23 and inhibits cytokine - cytokine receptor coupling and signaling
  Other Names: Stelara
Drug: Prednisone — Prednisone is an anti-inflammatory medication

SUMMARY:
The purpose of this study is to determine whether ustekinumab is effective in the treatment of Giant Cell Arteritis (GCA)

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of ustekinumab, an interleukin (IL)-12/23 inhibitor, in patients with GCA

Hypothesis IL-12/23 pathway blockade may maintain disease remission in patients with GCA

Specific Aims

* To evaluate the safety and tolerability of ustekinumab administration in 20 patients with GCA
* To evaluate the efficacy of ustekinumab for remission maintenance and glucocorticoid sparing in 20 patients with GCA

ELIGIBILITY:
Inclusion Criteria: Subjects must meet the following criteria

1. Able and willing to provide written informed consent and to comply with the study protocol
2. Diagnosis of GCA classified according to the following criteria:

   * Age 50 years or older
   * History of erythrosedimentation rate (ESR) ≥ 50 mm/hour or C-reactive protein (CRP) ≥ 10 mg/L

   AND at least one of the following:
   * Cranial symptoms of GCA
   * Symptoms of polymyalgia rheumatica (PMR)

   AND at least one of the following:
   * Temporal artery biopsy revealing features of GCA
   * Evidence of large-vessel vasculitis by angiography or cross-sectional imaging
3. Active new-onset or relapsing active disease

Exclusion Criteria:

1. Allergies: Subjects who have history of previous severe allergic or anaphylactic reaction associated with the administration of monoclonal antibodies or antibody fragments.
2. Systemic infection: Subjects who have an active systemic infection.
3. Serious infection: Subjects who have had serious infections, or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of enrollment.
4. Chronic or recurrent infection: Subjects who have chronic or recurrent bacterial, viral, fungal, mycobacterial, or protozoan infection.
5. Opportunistic infection: Subjects who have, or have had, an opportunistic infection within 6 months prior to enrollment.
6. Subjects who have active hepatitis B or active hepatitis C or a documented history of HIV
7. Latent tuberculosis infection
8. Malignancy
9. Subjects with evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, immunologic, psychiatric or gastrointestinal disease that could interfere with participation in the trial according to the protocol.
10. Subjects with transplanted organs (with the exception of a corneal transplant > 3 months prior to screening)
11. Major surgery within 8 weeks prior to Screening or planned major surgery within 12 months after Baseline
12. Pregnancy
13. The following laboratory abnormalities

    * Hemoglobin < 8 gr/dL
    * Platelets < 100/mm3
    * White blood cell count (WBC) < 3000/mm3
    * Absolute neutrophil count < 2000/mm3
    * Absolute lymphocyte count < 500/mm3
    * Serum creatinine > 1.4 mg/dL in female subjects and > 1.6 mg/dL in male subjects
    * Total bilirubin > 2 mg/dL
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 X upper limit of normal
    * Positive hepatitis B surface antigen, hepatitis B core antibody or hepatitis C antibody
14. Prohibited medications:

    * Subjects who received methotrexate (MTX) > 30 mg weekly, azathioprine, mycophenolate mofetil, cyclophosphamide, chlorambucil, tacrolimus, leflunomide, canakinumab, belimumab, abatacept, tocilizumab, secukinumab, infliximab, etanercept, adalimumab, golimumab, or certolizumab within the 3-month period prior to enrollment.
    * Subjects who had treatment with any anti-cluster designation antigen (CD)20 agent (e.g., rituximab) within the 9-month period prior to enrolment
    * Subjects who used any investigational drug within 1 month prior to enrollment or within 5 half-lives of the investigational agent, whichever is longer.
    * Low dose MTX: Patients on < 30 mg of MTX weekly will be eligible for enrollment after a 2-week washout interval before receiving ustekinumab
    * Vaccines: Subjects who received any live virus or bacterial vaccinations other than bacille Calmette-Guerin (BCG) within the 3 months before the first administration of the study agent, or are expected to receive any live virus or live bacterial vaccinations during the study, or up to 3 month after the last administration of ustekinumab are not eligible. Subjects who received BCG vaccines within the 12 months before the first administration of the study agent, or are expected to receive BCG vaccines during the study, or up to 12 month after the last administration of ustekinumab are also not eligible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Matza MA, Fernandes AD, Stone JH, Unizony SH. Ustekinumab for the Treatment of Giant Cell Arteritis. Arthritis Care Res (Hoboken). 2021 Jun;73(6):893-897. doi: 10.1002/acr.24200. PMID 32248659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2016 and August 2018, we screened 16 GCA patients for this trial. Three patients failed the screening process and 13 patients were enrolled.
Pre-assignment Details: Three patients failed the screening due to dementia (N = 1), severe prednisone-induced depression (N = 1), and positive hepatitis B core antibody (N = 1)
Groups:
- Ustekinumab Plus Prednisone: 1. Ustekinumab 90 mg was administered subcutaneously at baseline, week 4, week 12, week 20, week 28, week 36 and week 44.
     Ustekinumab: Ustekinumab is a humanized monoclonal antibody that targets the p40 subunit of IL-12 and IL-23 and inhibits cytokine - cytokine receptor coupling and signaling
  2. All patients received a 6 month prednisone course tapered according to predefined schedules starting at either 60 mg, 40 mg or 20 mg. The initial dose of prednisone was chosen by the investigators according to disease severity and comorbid medical conditions. The initial prednisone dose was 60 mg in 3 patients, 40 mg in 9 patients, and 20 mg in 1 patient.
  Prednisone is an anti-inflammatory medication
Period: Overall Study
Arm/Group | Ustekinumab Plus Prednisone
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ustekinumab Plus Prednisone: 1. Ustekinumab: 90 mg of ustekinumab will be administered subcutaneously at baseline, week 4, week 12, week 20, week 28, week 36 and week 44.
  2. Prednisone: All patients will receive a prednisone course tapered according to predefined schedules starting at either 60 mg, 40 mg or 20 mg. The initial dose of prednisone will be chosen by the investigators according to disease severity and comorbid medical conditions. The duration of the prednisone taper will be 6 months in all cases.
  Ustekinumab: Ustekinumab is a humanized monoclonal antibody that targets the p40 subunit of IL-12 and IL-23 and inhibits cytokine - cytokine receptor coupling and signaling
  Prednisone: Prednisone is an anti-inflammatory medication
Arm/Group | Ustekinumab Plus Prednisone
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Glucocorticoid-free Remission
Description: The primary study endpoint, prednisone-free remission, was defined as: 1) absence of relapse from the time that remission was achieved through week 52; 2) normalization of ESR (<40 mm/hour) and CRP (<10 mg/L); and, 3) adherence to the protocol prednisone taper.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Ustekinumab Plus Prednisone: 1. Ustekinumab 90 mg was administered subcutaneously at baseline, week 4, week 12, week 20, week 28, week 36 and week 44.
  2. All patients received a 6 month prednisone course tapered according to predefined schedules starting at either 60 mg (n = 3), 40 mg (n = 9) or 20 mg (n = 1).
Arm/Group | Ustekinumab Plus Prednisone
Number analyzed (Participants) | 13
Participants | 3

2. Secondary Outcome: Number of Participants With Disease Flare
Description: Disease relapse was defined as the recurrence of signs or symptoms of GCA (e.g., cranial or PMR) that required treatment intensification, regardless of the ESR and CRP levels.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ustekinumab Plus Prednisone
Number analyzed (Participants) | 13
Participants | 7

3. Secondary Outcome: Cumulative Prednisone Dose
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: mg of prednisone
Arm/Group | Ustekinumab Plus Prednisone
Number analyzed (Participants) | 13
mg of prednisone | 2289 (498)

4. Other Pre Specified Outcome: Number of Participants With at Least One Adverse Event
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ustekinumab Plus Prednisone
Number analyzed (Participants) | 13
Participants | 12

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | Ustekinumab Plus Prednisone
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab Plus Prednisone (N=13)
Diverticulitis (Gastrointestinal disorders) | 1 (1) — One patient developed mild diverticulitis, which was classified as a serious adverse event because it required hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab Plus Prednisone (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02955147/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02955147/ICF_001.pdf